CLINICAL TRIAL: NCT01226537
Title: Effect of Taurine on Glycemic Control in Type I and Type II Diabetic Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCT01225588; NCT01225588 (obsolete NCT alias)
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: it is a Group of Metabolic Diseases in; Which a Person Has High Blood Sugar, Either; Because the Body Does Not Produce Enough Insulin,; or Because Cells do Not Respond to the Insulin That; is Produced.
Keywords: Taurine,Diabetes mellitus,oxidative stress,glycemic control
MeSH Terms: interventions — Taurine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Diabetes Mellitus type 1 taurine (Active Comparator): A total of 20 patients with 10 Type I and 10 type II diabetic will be enrolled in the study.After the preliminary examinations, we will categorize 10 Type I and Type II patients into two groups randomly (each group contain 5 patients).500mg Taurine capsules will be given twice per day for 6 months.
  Interventions: Drug: Taurine
- Diabetes mellitus type 1 placebo (Placebo Comparator): A total of 20 patients with 10 Type I and 10 type II diabetic will be enrolled in the study.After the preliminary examinations, we will categorize 10 Type I and Type II patients into two groups randomly (each group contain 5 patients).500mg Taurine capsules will be given twice per day for 6 months.
  Interventions: Drug: Taurine
- Diabetes type 2 taurine (Active Comparator): A total of 20 patients with 10 Type I and 10 type II diabetic will be enrolled in the study.After the preliminary examinations, we will categorize 10 Type I and Type II patients into two groups randomly (each group contain 5 patients).500mg Taurine capsules will be given twice per day for 6 months.
  Interventions: Drug: Taurine
- Diabetes type 2 placebo (Placebo Comparator): A total of 20 patients with 10 Type I and 10 type II diabetic will be enrolled in the study.After the preliminary examinations, we will categorize 10 Type I and Type II patients into two groups randomly (each group contain 5 patients).500mg Taurine capsules will be given twice per day for 6 months.
  Interventions: Drug: Taurine

INTERVENTIONS:
Drug: Taurine — 500 mg taurine capsules twice per day for 6 months

SUMMARY:
Diabetes mellitus (DM) and its vascular complications are the one of the most prevalent diseases in the state of Qatar. It is a multifactorial disease associated with the development of retinopathy, nephropathy, neuropathy, cardiomyopathy, and severe vascular dysfunction. The complications of diabetes are caused by either insulin deficiency (type 1 DM) or insulin resistance (type II DM).Unfortunately, effective and sustainable prevention programs of diabetes are limited, and treatment options for type II DM are restricted. Current therapy is based upon control of blood glucose, cholesterol and triglycerides, primarily through insulin replacement in type I diabetes or oral hypoglycemic agents and/or insulin replacement in type II diabetes. New therapies able to prevent vascular complications of diabetes are needed to decrease the occurrence of end organ damage and improve the quality of life of the people. Safe and effective nutritional supplements that could be given along with the regular treatment of the patients that might reduce the need for insulin replacement therapy provide tighter glucose control and protect against oxidative stress and the vascular pathology associated with diabetes mellitus are the need of the hour. Our hypothesis is that supplementation of Taurine in the diets of diabetic patients might reduce the dose or need for insulin replacement therapy and protect them against oxidative stress that is responsible for the complications of diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Above 18-65 Years of old
3. Known diabetic patients with HbA1c>8.0%
4. People who provide signed informed consent -

Exclusion Criteria:

* 1. Pregnancy 2. Diabetic patients with HbA1c <8.0 % 3. Recent or prospective surgical interventions 4. Complications of Type I and Type II DM, e.g., Active cardiovascular disease, nephropathy, retinopathy, neuropathy 5. People who do not provide signed informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose 2) HbA1c 3) Lipid profile 4) Taurine 5) Insulin 6) Urine Micro albumin 7) Eye test | 9 months
  500mg Taurine capsules will be given twice per day for 6 months. After the medication, each month the following outcomes will be measured Fasting glucose 2) HbA1c 3) Lipid profile 4) Taurine 5) Insulin 6) Urine Micro albumin